CLINICAL TRIAL: NCT03369249
Title: Health and Justice: A Continuum of Care for HIV and SU for Justice-Involved Young Adults (PHASE 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Center for Court Innovation (Other); The National Center on Addiction and Substance Abuse at Columbia University (Other); National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Katherine Elkington, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7574; R01DA043122 (NIH)
Record Dates: First submitted 2017-11-30; First posted 2017-12-11 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: HIV/AIDS; HIV Infections; Substance Use; Substance Abuse; Substance Use Disorders; Sexually Transmitted Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Link2CARE (Experimental): This arm is comprised of participants randomized to the 4-session Link2CARE intervention.
  Interventions: Behavioral: Link2CARE
- Standard of Care (No Intervention): This arm is comprised of participants who will not receive the 4-session Link2CARE intervention.

INTERVENTIONS:
Behavioral: Link2CARE — The Link2CARE intervention consists of 4 sessions. Session 1 consists of a one-on-one meeting with a Health Coach, during which participants will be offered an oral rapid HIV test and STI test. Sessions 2, 3, and 4 are group-based. During these sessions, participants will engage in discussions and activities regarding sexual and substance use risk behaviors.
  Arms: Link2CARE

SUMMARY:
This research study proposes to embed HIV testing outreach workers from a young adult focused medical and HIV treatment program into an alternative sentencing program to deliver a new service delivery model (Link2CARE) that integrates evidence-based protocols for justice-involved young adults to: a) promote HIV and STI testing, and HIV and SU risk screening, b) provide onsite intervention, and c) cross-system linkage to HIV, STI, and SU care. Phase 1 has already been completed. In phase 1, the intervention components were adapted for use among justice involved young adults and the resulting protocols were piloted with justice involved young adults, finalizing the resulting 4-session Link2CARE intervention. In phase 2, we will test Link2CARE among N=450 justice-involved young adults enrolled at the alternative sentencing program and conduct process evaluations with N=15 alternative sentencing program staff.

ELIGIBILITY:
Young Adults

Inclusion Criteria:

* Between 18-24 years of age
* Currently enrolled at the alternative to sentencing program
* Conversant in English
* Engaged in any unprotected or vaginal sexual activity (in the past 12 months)

Exclusion Criteria:

* Cognitively unable to complete the interview
* HIV positive

Alternative to Sentencing Staff

Inclusion Criteria:

* Currently employed at the alternative to sentencing program
* Between ages of 18-80

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2017-12-09 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Elkington, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Kings County Criminal Court, Brooklyn, New York, United States

REFERENCES:
- [Derived] Ertl MM, Jones A, Hickson R, Achebe I, Gyamfi Ertl SL, Sichel CE, Campos S, O'Grady MA, Tross S, Wilson P, Cohall RM, Cohall AT, Elkington KS. Technology Access and Perceptions of Telehealth Services Among Young Adults Involved in the Court System. J Adolesc Health. 2024 Mar;74(3):582-590. doi: 10.1016/j.jadohealth.2023.09.019. Epub 2023 Dec 8. PMID 38069927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited at the County Court house; screening took place and if eligible the participant was scheduled an appointment for baseline survey and randomized to study group. The first session either happened the same day or a few days later if the participant was unable to stay following the survey
Groups:
- Standard of Care: This arm is comprised of participants who will not receive the 4-session Link2CARE intervention and instead receive services as usual.
Period: Overall Study
Arm/Group | Link2CARE | Standard of Care
Started | 152 | 155
Completed | 135 | 139
Not Completed | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Link2CARE | Standard of Care | Total
Number analyzed (Participants) | 152 | 155 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 155 | 307
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.23 (2.04) | 21.02 (2.08) | 21.13 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 111 | 118 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 11 | 13
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 100 | 103 | 203
  White | 8 | 11 | 19
  More than one race | 35 | 27 | 62
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 152 | 155 | 307

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Unprotected Anal and Vaginal Sex Occasions in Past 3 Months
Description: measured by participant report in the "Sexual Risk" section of the questionnaires
Time Frame: at 12-month follow-up
Measure: Mean (Standard Deviation); unit: unprotected sex occasions
Arm/Group | Link2CARE | Standard of Care
Number analyzed (Participants) | 152 | 155
unprotected sex occasions
  baseline | 32.76 (60.44) | 44.00 (76.65)
  12months | 27.70 (57.43) | 32.76 (73.37)
Statistical Analysis 1: Comparison: Link2CARE vs Standard of Care; Test type: Superiority; p = 0.635, generalized estimating equations — A priori threshold for statistical significance was <0.05; log ratio of rate ratios = 0.15, 95% CI 2-sided [-0.46 to 0.75], Standard Error of Mean 0.31 — Standard error of the Beta regression coefficient

2. Secondary Outcome: Frequency of Young Adults Substance Use in Past 30 Days
Description: measured by participant report in the "Substance Use" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

3. Secondary Outcome: Number of Young Adults Referred to Substance Use Treatment
Description: measured by Health Coach report in the Health Coach logs and participant report in the "Substance Use Referral" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

4. Secondary Outcome: Number of Young Adults Attending Intake Plus One Treatment Session
Description: measured by Health Coach report in the Health Coach logs and participant report in the "Substance Use Treatment" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

5. Secondary Outcome: Acceptance of STI Testing (Yes/no)
Description: measured by Health Coach report in the "Session 1 Sexual Risk" questionnaire
Time Frame: at day 1 of enrollment
Reporting Status: Not Posted

6. Secondary Outcome: Any STI Testing
Description: measured by participant report in the "STI Testing" section of the questionnaires
Time Frame: between 6- and 12-month follow-ups
Reporting Status: Not Posted

7. Secondary Outcome: Number of STI+ Young Adults Referred to STI Treatment
Description: measured by the Health Coach report in the Health Coach Logs and participant report in the "STI Referral" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

8. Secondary Outcome: Number of STI+ Young Adults Attending 1 or More Treatment Appointments
Description: measured by Health Coach report in the Health Coach logs and participant report in the "STI Treatment" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

9. Secondary Outcome: Acceptance of HIV Testing (Yes/no)
Description: measured by Health Coach report in the "Session 1 Sexual Risk" questionnaire
Time Frame: at day 1 of enrollment
Reporting Status: Not Posted

10. Secondary Outcome: Any HIV Testing
Description: measured by participant report in the "HIV Testing" section of the questionnaires
Time Frame: between 6-month and 12-month follow-ups
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of HIV+ Young Adults Referred to HIV Treatment
Description: measured by Health Coach report in the Health Coach logs and participant report in the "HIV Referral" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of HIV+ Young Adults Attending at Least One Treatment Appointment
Description: measured by Health Coach report in the Health Coach logs and participant report in the "HIV Treatment" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Number of Young Adults Behaviorally PrEP Eligible Referred to PrEP/Medical Care
Description: measured by Health Coach report in the Health Coach logs and participant report in the "PrEP Referral" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Number of Young Adults Behaviorally PrEP Eligible Attending at Least One HIV Care Appointment
Description: measured by Health Coach report in the Health Coach logs and participant report in the "PrEP Uptake" section of the questionnaires
Time Frame: at 3-, 6-, and 12-month follow-ups
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Link2CARE | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/152 | 1/155
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/155
Other Adverse Events (participants affected / at risk) | 24/152 | 25/155
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Link2CARE (N=152) | Standard of Care (N=155)
Suicidal Ideation (Social circumstances) | 24 | 25 — Assessed via beck depression inventory at each study interview (baseline, 3m, 6m and 12m)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (8):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/Prot_SAP_000.pdf
  • Informed Consent Form: Cover Sheet (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_001.pdf
  • Informed Consent Form: Authorization for the Release of Information (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_002.pdf
  • Informed Consent Form: YA IC for Participation in a Study BJI (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_003.pdf
  • Informed Consent Form: YA IC for Participation in a Study CASES (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_004.pdf
  • Informed Consent Form: HIPAA (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_005.pdf
  • Informed Consent Form: YA IC for HIV and/or STI Testing (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_006.pdf
  • Informed Consent Form: YA IC for HIV and/or STI Testing at 6 and12 Mo (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03369249/ICF_007.pdf